CLINICAL TRIAL: NCT05935787
Title: A Multicenter, Double-blind, Placebo-controlled, Randomized Study of the Efficacy and Safety of Sequential Therapy With CYTOFLAVIN® (NTFF POLYSAN, Russia), Solution for Intravenous Infusion and Enteric-coated Tablets, in the Complex Rehabilitation of Patients With Acute Stroke
Brief Title: Cytoflavin in the Complex Rehabilitation of Stroke Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: POLYSAN Scientific & Technological Pharmaceutical Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CTF-III-SR-2022
Record Dates: First submitted 2023-06-28; First posted 2023-07-07 (Actual); Last update posted 2025-08-15 (Actual); Status verified 2025-08

CONDITIONS: Stroke
Keywords: stroke rehabilitation
MeSH Terms: conditions — Stroke | interventions — cytoflavin; Inosine; Niacinamide; Riboflavin; Succinic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cytoflavin (Experimental)
  Interventions: Drug: Cytoflavin (Inosine + Nicotinamide + Riboflavin + Succinic Acid)
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Cytoflavin (Inosine + Nicotinamide + Riboflavin + Succinic Acid) — Cytoflavin (Inosine + Nicotinamide + Riboflavin + Succinic Acid), 20 ml (two ampoules of 10 ml each) once a day intravenously in a dilution of 200 ml of 0.9% sodium chloride solution at a rate 3-4 ml/min, for 15 days + Cytoflavin ((Inosine + Nicotinamide + Riboflavin + Succinic Acid), 2 tablets 2 times a day, for 25 days
  Arms: Cytoflavin
Drug: Placebo — Placebo, 20 ml (two ampoules of 10 ml each) once a day intravenously in a dilution of 200 ml of 0.9% sodium chloride solution at a rate 3-4 ml / min, for 15 days + Placebo, 2 tablets 2 times a day, for 25 days
  Arms: Placebo

SUMMARY:
It is known that the acute period of stroke occurs is accompanied by oxidative stress, when intense generation of reactive oxygen species (ROS) have a toxic effect, which causes oxidative degradation of proteins, lipids, nucleic acids. Antioxidants may have a positive effect on the processes of reparation, remodeling and neuroplasticity, thus improving the effectiveness of post-stroke rehabilitation. The adjunctive use of drug therapy that improves neuroplasticity may promote accelerated motor learning, which underlies the effects of exercise therapy and physical therapy, speech therapy, and sessions with a psychologist or occupational therapist. CYTOFLAVIN® is a combination of succinic acid, riboflavin, nicotinamide and inosine (riboxin) which has antihypoxic and antioxidant effects. The study hypothetizes that this neurometabolic drug will facilitate learning in stroke survivors and help to acquire new cognitive or motor skills necessary for daily living. The study will be conducted in two parallel groups of stroke survivors: the experimental group will be treated with Cytoflavin along with ohysical rehabilitation, the control group will receive standard rehabilitation course.

ELIGIBILITY:
Inclusion Criteria:

1. Signed Patient informed consent form
2. Men and women aged 40 to 80, inclusive.
3. Ischemic stroke in the carotid area, or hemorrhagic stroke in the cerebral hemispheres, occurred in the previous 14-90 days before screening.
4. Acute neuroimaging data (CT and/or MRI) do not contradict the clinical and topical diagnosis of stroke.
5. The presence of a measurable neurological deficit in the motor or sensory area.
6. Availability of rehabilitation potential, which is assessed by the specialists of the multidisciplinary team
7. Modified Rankin score 3-4.
8. The possibility to visit outpatient rehabilitation at the research center.
9. Ability to understand and comply with protocol requirements.
10. For women: consent to use reliable methods of contraception or absent reproductive potential.
11. For men: consent to the use of adequate methods of contraception, or complete abstinence from sexual activity for the period of the study, or absent reproductive potential.

Exclusion Criteria:

1. Known hypersensitivity to any component of the study drug
2. Severe visual and hearing impairments that prevent the implementation of study procedures.
3. Severe spasticity (scored 3-4 by Ashworth scale).
4. Impaired swallowing, which does not allow taking drugs orally.
5. Communication deficit that does not allow the patient to fulfill the conditions of the study protocol (including total aphasia).
6. The presence of contraindications to complex rehabilitation in a hospital (lack of rehabilitation potential, somatic diseases that prevent a complex of rehabilitation measures).
7. Aneurysmal subarachnoid hemorrhage.
8. Previous (before the actual ictus) stroke with residual neurological deficit.
9. Disability is primarily not attributed to the last stroke
10. Severe renal failure
11. Severe liver failure
12. End stage of other chronic incurable diseases.
13. Decompensated diabetes mellitus.
14. History of cancer, mental illness, HIV infection, syphilis, tuberculosis, alcohol, drug or drug addiction.
15. Established diagnosis of a mental or neurodegenerative disease
16. Constant use of psychotropic drugs (neuroleptics, tranquilizers, antidepressants) or nootropic drugs in the previous 3 months before the patient was included in the study, except for stroke treatment in acute hospital.
17. Alcohol or drug addiction

19. Pregnancy, lactation.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Actual)
Dates: Start 2023-06-09 (Actual); Primary Completion 2024-08-01 (Actual); Study Completion 2024-12-07 (Actual)

PRIMARY OUTCOMES:
Change of performance | 40 days
  Change at the performance subscale (range 0-10, higher=better) of Canadian Occupational Performance Measure (COPM) score after completion of therapy compared to baseline

CONTACTS AND LOCATIONS:
Overall Officials: Alexey Shmonin, Prof, Study Director — First St. Petersburg State Medical University named after I.P. Pavlov
Locations (3):
- Russia (3):
  - City General Hospital №2, Saint Petersburg
  - City Hospital №40 of the Kurortny District, Saint Petersburg
  - Saint-Petersburg I.I.Dzanelidze Research Institute of Emergency Medicine, Saint Petersburg

IPD SHARING:
Plan to Share IPD: No